CLINICAL TRIAL: NCT01428037
Title: A Randomized,Double-blind,Placebo-controlled, Multicenter Study of the Efficacy and Safety of Vaginal Misoprostol for Cervical Ripening and Induction of Labor
Brief Title: Safety and Efficacy Study of Vaginal Misoprostol for Cervical Ripening and Induction of Labor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regenex Pharmaceutical, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RH-MS-01RCT
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Cervical Ripening; Induction of Labor
Keywords: Vaginal Misoprostol; Cervical Ripening; Labor Induced

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol Vagianl Tablet (Experimental): Misoprostol Vaginal Tablet 25 mcg.
  Interventions: Drug: Misoprostol vaginal Tablet 25 mcg
- Placebo (Placebo Comparator): Tablet without active ingredient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — One tablet vaginal inserted at 4 hrly interval with maximum of three doses
  Arms: Placebo
Drug: Misoprostol vaginal Tablet 25 mcg — One tablet vaginal insert at 4 hrly interval with maximum of three doses
  Other Names: Misoprostol vaginal Tablet
  Arms: Misoprostol Vagianl Tablet

SUMMARY:
The purpose of this study is to estimate the efficacy and safety of the 25mcg vaginal misoprostol for cervical ripening and induction of labour.

DETAILED DESCRIPTION:
There are many pregnant women require medical intervention to induce labor for some reasons at term. There are two fundamental changes that characterize pre-labor preparation for delivery: sensitization of the myometrium to produce contractions, and ripening (softening and dilation) of the cervix. A synthetic Prostaglandin misoprostol is fundamental to both of these changes. Low dose misoprostol is effective and safe for labor induction and has been used widely.

Oral tablets(200mcg) are broken into fragments and used intravaginally to ripen the cervix and induce labor due to the disadvantages of existing cervical ripeners (delivery of bolus doses, freezer or refrigerated storage, lack of efficacy in labor induction), and due to safety concerns with the off-label use of oral misoprostol tablet fragments, Regenex Corporation has developed a vaginal tablet with 25mcg misoprostol.

The primary objective of the study was to assess of the efficacy and safety of low dose (25 mcg) of misoprostol vaginal tablet for cervical ripening and induction of labour.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Aged 20 years or older.
* At term (37 to 42 weeks inclusive gestation).
* Cephalic presentation (normal lie).
* No rupture.
* Bishop score ≤6.
* With an indication for labour induction.
* Written informed consent.

Exclusion Criteria:

* Any contraindication to vaginal delivery.
* Previous of uterine scar(Cesarean section or other uterine surgeries).
* Heavy or repeated vaginal bleeding in third trimester of pregnancy.
* Have a history of glaucoma,asthma or epilepsy.
* Contraindication to prostaglandin use.
* Known severe allergy to prostaglandin.
* Placenta previa
* Premature rupture of membranes
* Placental abruption
* Fetal malpresentation(Breech or Transverse)
* Obvious cephalopelvic disproportion
* Amniotic Fluid Index more than 250mm or less than 50mm
* Fetal growth restriction
* Fetal malformation
* Fetal distress
* Preeclampsia or eclampsia
* Fetal macrosomia of prenatal diagnosis(B-type ultrasonic inspection/Abdomen estimates)
* Intrahepatic cholestasis syndrome(ICP)
* Pregnancy with severe heart, lung, liver, kidney, endocrine disease and immune dysfunction
* Pregnancy with acute systemic infection
* Pregnancy with Severe anemia
* Cervical carcinoma
* Some genital tract infection disease, such as active herpes infection
* Take part in other clinical trials within three months.
* The person that investigator thought not be enrolled.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Treatment success rate | From the first dose to 12-24 hours
  Treatment success is defined as: ≧3 of Bishop score increased within 12 hours or Vaginal delivery within 24 hours.

SECONDARY OUTCOMES:
Percentage of participants of labor onset within 24 hours | From the first dose to 24 hours
Time from 1st dose to labor onset | From the first dose to labor onset
Need for augmentation of labor with oxytocin | From the first dose to neonate delivery
Rate and reason for Cesarean Section | From the first dose to neonate delivery

CONTACTS AND LOCATIONS:
Overall Officials: Wen Di, MD, Principal Investigator — RenJi Hospital
Locations (6):
- China (6):
  - Zhongda Hospital ,Southeast University, Nanjing, Jiangsu
  - The First Affliated Hospital with Nanjing Meical Uniersity, Nanjing, Jiangsu
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Southwest Hospital, Chongqing
  - The International Peace Maternity & Child Care of China Welfare Institute, Shanghai
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai